CLINICAL TRIAL: NCT02994316
Title: Interest of Plasma Copeptin Levels in Management of Children With Diabetic Ketoacidosis
Brief Title: Plasma Copeptin Levels in Children With Diabetic Ketoacidosis
Acronym: COPACD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9649
Record Dates: First submitted 2016-11-28; First posted 2016-12-15 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Diabetic Ketoacidosis Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- children under the age of 16 diabete with ketoacidosis (Experimental): At diagnosis mellitus type 1 (measure of blood glucose level) bicarbonate levels will be measured and children will included in the arm "with ketoacidosis (bicarbonate < 15mmol/L)
  Interventions: Other: Copeptine dosage in children with diabetic ketoacidosis at diagnosis
- children under the age of 16 diabete without ketoacidosis (Sham Comparator): At diagnosis mellitus type 1 (measure of blood glucose level) bicarbonate levels will be measured and children will included in the arm "without ketoacodosis (bicarbonate> 15 mmol/L)
  Interventions: Other: Copeptine dosage in children with diabetic ketoacidosis at diagnosis

INTERVENTIONS:
Other: Copeptine dosage in children with diabetic ketoacidosis at diagnosis — Blood collection of 3 mL for copeptin dosage will be taken at different times in the first hours of management of diabetic ketoacodosis in children under the age of 16 years

SUMMARY:
Children with diabetic ketoacidosis risk neurological complications such as cerebral edema with high morbidity. To prevent cerebral edema, it is essential to control correction of hypovolemia, hyperglycemia and natremia. Markers usually used in management of diabetic ketoacidosis don't always permit an optimal care.

Plasma copeptin levels reflect vasopressin secretion which is high in diabetic ketoacidosis.

Therefore, monitoring of plasma copeptin levels could be of interest in children with diabetic ketoacidosis and risk of sévère neurological complications.

DETAILED DESCRIPTION:
Biological risk factors for severe complications in diabetic ketoacidosis are described (high blood glucose level, metabolic acidosis, high blood urea nitrogen, hypernatremia) but their dosage and monitoring are not sufficient to distinguish high risks situations.

Several studies suggest that vasopressin secretion is increased in diabetic ketoacidosis. This high level could be important in occurrence of cerebral edema. Monitoring of vasopressin levels could then have an interest in patients at risk of severe complications but reliability of copeptin dosage depend of collection conditions and its packaging. These conditions are difficult to ensure and copeptin dosage, which represent vasopressin secretion, is easier to perform.

Copeptin dosage could then be a new biological marker, more accurate and specific, for an optimal management of diabetic ketoacidosis.

This type of study has never been carried out neither in children nor in adults.

ELIGIBILITY:
Inclusion criteria:

* Children between 6 months and 16 years
* Diagnosis of diabetes mellitus type 1 (cardinal syndrome, blood glucose level > 7 mmol/L in the fasted state or > 11 mmol/L not in fasted state, no signs for another type of diabetes mellitus)
* Children who need an exclusive intravenous rehydration for 36 hours
* Written informed consent of legal representative and of the child if possible
* Beneficiary of State Social Insurance

Exclusion criteria:

* Child under the age of 6 months or older than 16 years
* Non exclusive intravenous réhydration for at least 36 hours
* Child moved from another institution and for whom an intravenous rehydration or insulin therapy have already begun
* Non type 1 diabetes mellitus
* Non affiliation to State Social Insurance

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Interest of copeptin dosage as a severity marker in children under the age of 16 with diabatic ketoacidosis | 36 hours
  Study of correlation between copeptin levels and metabolic acidosis management of diabatic ketoacidosis in children

SECONDARY OUTCOMES:
Correlation between plasma copeptin levels and other markers used in management of diabatic ketoacidosis in the first 36 hours after diagnosis- Plasma copeptin levels at diagnosis of diabate mellitus type 1 without ketoacidosis in children | 36 hours
  Interest of copeptin dosage as a new marker of diabatic ketoacidosis severy compared to other used markers

CONTACTS AND LOCATIONS:
Overall Officials: GILLES GC CAMBONIE, PU PH, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No